CLINICAL TRIAL: NCT05902624
Title: Evaluation of the Efficacy of Cryotherapy Combined With Intralesional Hepatitis B Virus Vaccine Versus Either Therapy in the Treatment of Multiple Cutaneous Warts :a Comparative Study
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maria Awny Armia, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cutaneous warts treatment
Record Dates: First submitted 2023-04-03; First posted 2023-06-15 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Cutaneous Warts
MeSH Terms: interventions — Hepatitis B Vaccines; Cryotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group intralesional injection of HBV vaccine (Other): Group 1: will include 20 patients with multiple cutaneous warts. They will be treated by intralesional injection of HBV vaccine into the largest wart by an insulin syringe every 2-weeks until complete clearance or for a maximum of 5 sessions.
  Interventions: Drug: Hepatitis B Virus Vaccine(HBV)
- Group cryotherapy (Other): Group 2: will include 20 patients with multiple cutaneous warts. They will be treated by cryotherapy every 2-weeks until complete clearance or for a maximum of 5 sessions.
  Interventions: Drug: Hepatitis B Virus Vaccine(HBV)
- Group cryotherapy with intralesional injection of HBV vaccine (Other): Group 3: will include 20 patients with multiple cutaneous warts. They will be treated by cryotherapy with intralesional injection of HBV vaccine into the largest wart by an insulin syringe every 2-weeks until complete clearance or for a maximum of 5 sessions.
  Interventions: Drug: Hepatitis B Virus Vaccine(HBV)

INTERVENTIONS:
Drug: Hepatitis B Virus Vaccine(HBV) — Hepatitis B Virus Vaccine(HBV)
  Other Names: cryotherapy

SUMMARY:
1. investigate the efficacy and safety of combined cryotherapy with intralesional HBV vaccine injection in the treatment of multiple common warts.
2. compare the efficacy and safety of the combined treatment versus either therapy in the treatment of multiple cutaneous warts.

DETAILED DESCRIPTION:
Introduction:

Warts are common, benign and epithelial proliferations and growths affecting the skin and/or the mucosa (Sterling JC,et al.,2014) caused by human papilloma virus (HPV) which is a double stranded DNA virus with a worldwide distribution(Pérez-González et al., 2022).

There are approximately 218 types of HPV identified as causing infections in humans (Magalhães et al., 2021).

Infection occurs predominantly via direct contact, although skin lesions can be transmitted indirectly, via contaminated surfaces, Abrasions and microtraumas expose the basal layer keratinocytes and facilitate contagion (EgawaN,et al 2015 and Vlahovic T.C.et al,2016).

The clinical manifestations of HPV-related diseases vary depending upon the HPV type and the site of inoculation (Burlamaqui et al., 2017).Extragenital cutaneous warts can present as common warts, plane warts, plantar warts (Abeck D. et al, 2019).HPV infection is one of the most common sexually transmitted infections with the most common manifestation of HPV in the genital area is anogenital warts or condylomata acuminate (Gofur, 2022). Infections due to these viruses may result in a wide spectrum of clinical manifestations in the skin and mucosa(Cubie, 2013).

Although cutaneous warts are mostly benign with spontaneous resolution after months or years in healthy patients, (Mohammed et al., 2022). Nonetheless, they can grow, cause discomfort or embarrassment to patients, or persist for months or years, increasing viral transmission between individuals. Also, anogenital warts caused by high risk strains possess an oncogenic potential (Magalhães et al., 2021).

Several therapeutic modalities have been used to treat HPV infections. The choice of treatment should take into account factors such as age, location, number and size of the lesions, clinical subtype and the patient's immunological status.(Araújo et al., 2021) Available treatment modalities include physical destruction (e.g., cryotherapy, electrosurgery, ablative laser, or surgical removal), chemical destruction (e.g., salicylic acid or trichloroacetic acid), and anti-proliferative agents (e.g., podophyllin, 5-fluorouracil or bleomycin). Unfortunately, no treatment has yet shown 100% effectiveness as a cure. Furthermore these modalities have side-effects (e.g. pain, erythema, burning sensation and scarring) (Ockenfels HM. 2016 and Ju et al, 2022) .Classical treatment lines are associated with high recurrence rates as they are limited to local application and do not act systemically (Raghukumar S et al 2017).So, there is a need for therapies with a greater efficacy and minimal side-effects ( Sterling JC,et al 2014).

Cryocautery represents a first line of therapy for cutaneous warts. It uses liquid nitrogen to freeze tissues and destroy warts (4).

Liquid nitrogen cryotherapy involves freezing a wart with liquid nitrogen for 10 to 20 seconds every two to three weeks. Precisely how cryotherapy destroys warts is not well understood, but the prevailing theory is that freezing causes local irritation, leading the host to mount an immune reaction against the virus (5) Immunotherapeutic agents act by enhancing the host cell-mediated immunity that helps to eliminate the virus rather than simply destroying visible skin lesions and have recently received increasing attention for the treatment of warts because of their non-destructive action, high safety profiles, promising results, and low recurrence rates. Contact immunotherapy using contact sensitizers (diphenylcyclopropenone or dinitrochlorobenzene), topical imiquimod, oral cimetidine or intralesional immunotherapy has been attempted as viable immunotherapeutic options for treatment of warts. (Ju et al., 2022).

Intralesional immunotherapy has been assessed as an alternative therapeutic approach, particularly for cases of recalcitrant or multiple warts, since it may facilitate the clearance of not only the injected wart but also surrounding non-injected warts. Various immunotherapeutic agents including skin test antigens (mumps, Candida, and Trichophyton); the combined measles, mumps, and rubella vaccine(MMR); the tuberculin purified protein derivative(PPD); Mycobacterium w vaccine; and bacillus Calmette-Guérin(BCG) vaccine have been assessed(Thappa DM, et al, 2016 ) (Ju et al., 2022).

Hepatitis B virus (HBV) vaccine is a highly safe and effective DNA vaccine against HBV infection that is recommended for all infants at birth and for children. It is also recommended for adults at high risk for infection because of their jobs, lifestyle, or living situations. It is relatively cheap, easy to produce, and extremely stable. Besides, HBV vaccination is associated with the stimulation, not only of humoral immunity that induces antibody production against Hepatitis B surface antigen (HBsAg), but also of cell-mediated immunity, particularly T helper1 Th1 cytokines such as interferon γ( IFN-γ )and interleukin2(IL-2). Furthermore, HBV vaccine has the advantage of being a non-live vaccine that can be used safely in immunocompromised patients in contrast to the live vaccines such as measles, mumps, and rubella (MMR), Bacillus Calmette-Guerin (BCG) that may pose high risks to the immunocompromised patients (Huang QD,et al. 2018).

Only two researches studied the efficacy of intralesional HBV vaccine injection in treatment of multiple common warts (Nofal et al., 2021, Nofal et al., 2022). Both studies revealed low success rate (20.7% and 23.3% respectively) of intralesional HBV vaccine at a dose of 0.2ml injected into the largest wart in biweekly sessions for a maximum of 5 sessions. It Worth mentioning that one the two studies also examined the efficacy of intramuscular injection of HBV vaccine at higher doses (0.5 ml and 1 ml/ injection) for 3 injections and reported a complete clearance of common warts in 50% of the patients, which was statistically significant higher than percentage of those patients who achieved complete clearance after treatment with intralesional injection of HBV vaccine using 0.2 ml/session for five sessions(Nofal et al., 2022). Whether this significant difference is related to the different treatment dosage or to the different administration routes is still to be unraveled by further studies.

ELIGIBILITY:
Inclusion Criteria:

* Any patients with multiple cutaneous warts of any site.
* Patients age above 10 years old
* No concurrent systemic or topical treatment of warts

Exclusion Criteria:

* Pregnancy and lactation.
* History of any bleeding, clotting disorder or using anticoagulants
* Chronic systemic diseases such as chronic renal failure, hepatic insufficiency, and cardiovascular disorders.
* Concurrent use of systemic or topical treatments of warts.
* Patients with history of neuropathy or peripheral ischemia.
* Patients with signs of inflammation or infection.
* Patients with history of a serious systemic or anaphylactic reaction or allergy to a prior dose of HBV vaccine or to any of its components.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Investigate the efficacy and safety of combined cryotherapy with intralesional HBV vaccine injection in the treatment of multiple common warts. | 10 weeks
  size of cutaneous warts in millimeters will be measured every visit
Compare the efficacy and safety of the combined treatment versus either therapy in the treatment of multiple cutaneous warts. | 10 weeks
  number of cutaneous warts will be measured every visit

CONTACTS AND LOCATIONS:
Overall Officials: Maria Awny, Master, Principal Investigator — Assiut University

REFERENCES:
- [Background] Nofal A, Salah E, Nofal E, Yosef A. Intralesional antigen immunotherapy for the treatment of warts: current concepts and future prospects. Am J Clin Dermatol. 2013 Aug;14(4):253-60. doi: 10.1007/s40257-013-0018-8. PMID 23813361
- [Background] Thappa DM, Chiramel MJ. Evolving role of immunotherapy in the treatment of refractory warts. Indian Dermatol Online J. 2016 Sep-Oct;7(5):364-370. doi: 10.4103/2229-5178.190487. PMID 27730031
- [Background] Araujo MG, Magalhaes GM, Garcia LC, Vieira EC, Carvalho-Leite MLR, Guedes ACM. Update on human papillomavirus - Part II: complementary diagnosis, treatment and prophylaxis. An Bras Dermatol. 2021 Mar-Apr;96(2):125-138. doi: 10.1016/j.abd.2020.11.005. Epub 2021 Feb 16. PMID 33637397
- [Background] Burlamaqui JC, Cassanti AC, Borim GB, Damrose E, Villa LL, Silva L. Human Papillomavirus and students in Brazil: an assessment of knowledge of a common infection - preliminary report. Braz J Otorhinolaryngol. 2017 Mar-Apr;83(2):120-125. doi: 10.1016/j.bjorl.2016.02.006. Epub 2016 Apr 22. PMID 27170346
- [Background] Mohammed GF, Al-Dhubaibi MS, Bahaj SS, Elneam AIA. Systemic immunotherapy for the treatment of warts: A literature review. J Cosmet Dermatol. 2022 Nov;21(11):5532-5536. doi: 10.1111/jocd.15330. Epub 2022 Aug 31. PMID 36017650
- [Background] Nofal A, Elaraby A, Elkholy BM. Intralesional Versus Intramuscular Hepatitis B Virus Vaccine in the Treatment of Multiple Common Warts. Dermatol Surg. 2022 Nov 1;48(11):1178-1184. doi: 10.1097/DSS.0000000000003595. Epub 2022 Sep 23. PMID 36165681
- [Background] Nofal A, Elsayed E, Abdelshafy AS. Hepatitis B virus vaccine: A potential therapeutic alternative for the treatment of warts. J Am Acad Dermatol. 2021 Jan;84(1):212-213. doi: 10.1016/j.jaad.2020.04.128. Epub 2020 Apr 29. No abstract available. PMID 32360758
- [Background] Perez-Gonzalez A, Cachay E, Ocampo A, Poveda E. Update on the Epidemiological Features and Clinical Implications of Human Papillomavirus Infection (HPV) and Human Immunodeficiency Virus (HIV) Coinfection. Microorganisms. 2022 May 18;10(5):1047. doi: 10.3390/microorganisms10051047. PMID 35630489
- [Background] Colpani V, Soares Falcetta F, Bacelo Bidinotto A, Kops NL, Falavigna M, Serpa Hammes L, Schwartz Benzaken A, Kalume Maranhao AG, Domingues CMAS, Wendland EM. Prevalence of human papillomavirus (HPV) in Brazil: A systematic review and meta-analysis. PLoS One. 2020 Feb 21;15(2):e0229154. doi: 10.1371/journal.pone.0229154. eCollection 2020. PMID 32084177
- [Background] Abou-Taleb DAE, Abou-Taleb HA, El-Badawy O, Ahmed AO, Thabiet Hassan AE, Awad SM. Intralesional vitamin D3 versus intralesional purified protein derivative in treatment of multiple warts: A comparative clinical and immunological study. Dermatol Ther. 2019 Sep;32(5):e13034. doi: 10.1111/dth.13034. Epub 2019 Aug 7. PMID 31355514
- [Background] Magalhaes GM, Vieira EC, Garcia LC, De Carvalho-Leite MLR, Guedes ACM, Araujo MG. Update on human papilloma virus - part I: epidemiology, pathogenesis, and clinical spectrum. An Bras Dermatol. 2021 Jan-Feb;96(1):1-16. doi: 10.1016/j.abd.2020.11.003. Epub 2020 Dec 10. PMID 33341319
- [Background] Ju HJ, Park HR, Kim JY, Kim GM, Bae JM, Lee JH. Intralesional immunotherapy for non-genital warts: A systematic review and meta-analysis. Indian J Dermatol Venereol Leprol. 2022 Nov-Dec;88(6):724-737. doi: 10.25259/IJDVL_1369_20. PMID 35962514
- [Background] Cubie HA. Diseases associated with human papillomavirus infection. Virology. 2013 Oct;445(1-2):21-34. doi: 10.1016/j.virol.2013.06.007. Epub 2013 Aug 9. PMID 23932731